CLINICAL TRIAL: NCT03530488
Title: The Value of Endocervical and Endometrial Lidocaine Flushing Before Office Hystroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pain During Hystroscopy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine group (Active Comparator): intrauterine and intracervical instillation of 4 ml of lidocaine 2% diluted in 15 ml normal saline 5 minutes before hystroscopy
  Interventions: Drug: Lidocaine; Procedure: Office hystroscopy
- control group (Placebo Comparator): intrauterine and intracervical instillation of 19 ml normal saline 5 minutes before hystroscopy
  Interventions: Procedure: Office hystroscopy

INTERVENTIONS:
Drug: Lidocaine — intrauterine and intracervical instillation of 4 ml of lidocaine 2% diluted in 15 ml normal saline
  Arms: Lidocaine group
Procedure: Office hystroscopy — A rigid 3.5 mm hystroscope with an optic of 30 degrees was used. Normal saline solution was used as distension media, with 120 mmHg intrauterine pressure, Vaginoscopic approach, nocervical tenaculum or dilators used.

SUMMARY:
women candidate for office hystroscopy were randomized to either flushing of the endocervix and endometrium with 4 ml lidocaine 2% diluted in 15 ml normal saline or 19 ml normal saline before office hystroscopy

DETAILED DESCRIPTION:
Patients were asked to urinate to evacuate the bladder. Posterior vaginal retractor was introduced to expose the cervix and ( embryo transfer catheter was introduced throught the cervix passing the internal os and intrauterine and intracervical instillation of to either flushing of the endocervix and endometrium with 4 ml lidocaine 2% diluted in 15 ml normal saline or 19 ml normal saline.

After 5 mins the procedure was started A rigid 3.5 mm hystroscope with an optic of 30 degrees was used. Normal saline solution was used as distension media, with 120 mmHg intrauterine pressure, Vaginoscopic approach, nocervical tenaculum or dilators used.

Post procedure pain management by optional dose of 75 mg of diclofenac potassium when requested.

ELIGIBILITY:
Inclusion Criteria:

* all women indicated for office hysteroscopy for evaluation of the uterine cavity eg: AUB, infertility

Exclusion Criteria:

* Women allergic to local anesthesia those required operative hysteroscopy under general anesthesia pelvic inflammatory disease known cervical malignancy profuse uterine bleeding, marked cervical stenosis recent uterine perforation previous cervical surgery and neurological disorders affecting evaluation of pain using other products that could affect the consistency of the cervix such as local estrogen, misoprostol or laminaire are contraindications for office hystroscopy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain assessment during the hysteroscopy | during hystroscopy procedure
  pain assessment during hystroscopy using visual analogue scale VAS. is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100

SECONDARY OUTCOMES:
Pain assessment 10 minutes after hysteroscopy | 10 minutes after hysteroscopy
  pain assessment 10 minutes after hystroscopy using visual analogue scale VAS. is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100
Pain assessment 30 minutes after hysteroscopy | 30 minutes after hysteroscopy
  pain assessment 30 minutes after hystroscopy using visual analogue scale VAS. is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100
Pain assessment 60 minutes after hysteroscopy | 60 minutes after hysteroscopy
  pain assessment 60 minutes after hystroscopy using visual analogue scale VAS. is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shoab AY, Maged AM, Ramadan W, Dahab S, Deeb WS, Ali YZA, Mostafa WAI, Hussein EA. The value of endocervical and endometrial lidocaine flushing before office hysteroscopy: A randomized controlled trial. Int J Gynaecol Obstet. 2020 Jan;148(1):113-117. doi: 10.1002/ijgo.12992. Epub 2019 Oct 19. PMID 31593299